CLINICAL TRIAL: NCT00592423
Title: Effect of Neck Rotation and Continuous Positive Airway Pressure (CPAP) on Upper Airway Anatomy in Anesthetized Children - an MRI Study
Brief Title: CPAP and Lateral Neck Rotation on Anesthetized Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary data was inconclusive to warrant keeping the study open.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Ronald Litman, DO,, The Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004-10-3977
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Hypoventilation
Keywords: Lateral neck rotation; Continuous Positive Airway Pressure
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): A "convenience" sample of children will be utilized for this study, which will include both genders and all ethnicities. There is no known predilection for any racial or gender inequalities with regard to subject recruitment or outcome variables related to this study.
  Interventions: Other: Continuous Positive Airway Pressure during MRI

INTERVENTIONS:
Other: Continuous Positive Airway Pressure during MRI — 10 cm H20 pressure for CPAP while lateral neck positioning is done for MRI - each side should take 5 minutes.

SUMMARY:
The primary aim of this study is to determine the changes in upper airway anatomy that occur during lateral neck rotation and subsequent administration of continuous positive airway pressure (CPAP) in anesthetized, spontaneously breathing children. The hypothesis for this study is that neck rotation decreases overall upper airway volume because of constriction at the level of the larynx, and that this constriction is relieved by administration of CPAP.

DETAILED DESCRIPTION:
The most commonly performed surgical procedure requiring general anesthesia in the pediatric population is myringotomy and placement of pressure equalizing tubes in the middle ear. It is performed in otherwise healthy children with chronic middle ear fluid collections and infections. In these cases, general anesthesia is accomplished by inhalation of a volatile anesthetic gas, which induces unconsciousness and analgesia for the approximately 10 minutes it takes to perform the procedure. A requirement of the procedure is lateral neck rotation by the anesthesiologist managing the airway. This enhances surgical visibility (Fig 1). However, a well-known clinical consequence of lateral neck rotation is development of upper airway obstruction with subsequent hypoxemia.1 Anesthesiologists routinely counteract this problem by placement of an oral airway device or application of CPAP, or both. Nevertheless, intervening hypoxia often necessitates temporary halting of the procedure and resumption of the neutral neck position until hypoxemia abates. This study will determine the anatomical mechanism for upper airway obstruction during lateral neck rotation and will elucidate the effects of administration of CPAP on this obstruction.

This study will use an MRI imaging technique that has been used recently at CHOP by Drs. Raanan Arens and Soroosh Mahboubi to study the three-dimensional characteristics of the upper airway in children. This methodology, which was developed at the University of Pennsylvania and CHOP, utilizes fuzzy connectedness-based automatic segmentation that allows visualization of the upper airway in a correct anatomical orientation as it relates to airflow.2,3 This technology has been successfully applied to anesthetized children without any apparent adverse effects (see IRB # 2003-2-3189).

An additional evaluable patient will be photographed during elective bronchoscopy with general anesthesia to correlate the MRI images with images visualized clinically.

ELIGIBILITY:
Inclusion Criteria:

1. MRI: Children requiring MRI examination with propofol sedation.
2. Bronchoscopy: Child requiring elective flexible bronchoscopy during general anesthesia. (1 child only) -

Exclusion Criteria:

1. Acute or chronic lung disease,
2. upper airway disease,
3. congestive heart failure,
4. obesity,
5. sleep apnea syndrome,
6. central nervous system disease likely to influence muscle tone,
7. any type of abnormality in head or neck anatomy, or
8. the requirement for any type of airway adjunct device (e.g., oral airway, endotracheal tube, etc.). -

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2005-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
This study will determine the anatomical mechanism for upper airway obstruction during lateral neck rotation and will elucidate the effects of administration of CPAP on this obstruction. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Litman, DO, Principal Investigator — Children's Hospital of Philadelphia